CLINICAL TRIAL: NCT04931758
Title: Validation of the French Version of the Fremantle Back Awareness Questionnaire (FreBAQ) in Patients With Chronic Low Back Pain
Acronym: FreBAQ
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2020-2/AH-1; 2021-A00373-38 (Other: ANSM)
Record Dates: First submitted 2021-06-03; First posted 2021-06-18 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with low back pain
  Interventions: Other: Pain Questionnaire
- Controls
  Interventions: Other: Pain Questionnaire

INTERVENTIONS:
Other: Pain Questionnaire — Subjects will take the FreBAQ questionnaire at Day 0 and a subgroup of 35 controls and 15 patients will take the same questionnaire at Day 7

SUMMARY:
In patients with chronic low back pain, the Fremantle Back Awareness Questionnaire (FreBAQ) measures the duration and intensity of pain and functional limitations. The FreBAQ is a simple tool created to assess disturbances in the body representation of the back, and the only one existing in chronic low back pain. It is a 9-item self-questionnaire in which each item is measured on a 5-point Likert scale ranging from "Never (score of 0)" to "Always (score of 4)". It assesses neglect, perceived body image of the back, accuracy in proprioceptive perception of back movements.

The psychometric properties of the FreBAQ in English, Japanese, Dutch, Turkish and German are validated and acceptable; however, they have never been studied in French and no validated version of this questionnaire in French exists.

The study investigators hypothesize that the French version of the FreBAQ has good psychometric qualities, allowing it to be used in the French chronic low back pain population.

ELIGIBILITY:
Inclusion Criteria:

* Subject with no history of chronic low back pain and with a lumbar VAS <2 for more than 3 months.
* Patient with chronic low back pain: pain localized between the edge of the last lower ribs and the intergluteal groove (17) for more than 3 months.
* Patient with a lumbar VAS > 2 for more than 3 months.
* Patient whose low back pain is of common origin (no underlying organic etiology).
* In case of lumbar-radicular pain, patient with a VAS (lumbar) > VAS (leg)
* Patient who speaks and understands French
* Patient with no history of arthrodesis or lumbar disc prosthesis
* Subject affiliated or beneficiary of a health insurance plan.
* The patient must have given their free and informed consent and signed the consent form

Exclusion Criteria:

* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Patient pregnant, parturient or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic low back pain defined as pain localized between the edge of the last lower ribs and the intergluteal groove (17) for more than 3 months followed in the Physical Medicine and Rehabilitation Department of the CHU of Nîmes and persons recruited among the members of the service and their entourage, as well as all patients coming for consultation in the service with no history of chronic low back pain and lumbar VAS < 2 for more than 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Pre-test of French version of FreBAQ on 20 representative patients | Baseline
  9-item self-administered questionnaire newly translated into French using a standard translation-retro-translation system, each item measured on a 5-point Likert scale ranging from "Never (score of 0)" to "Always (score of 4)

SECONDARY OUTCOMES:
FreBAQ score | Day 0
  a 9-item self-administered questionnaire, each item measured on a 5-point Likert scale ranging from "Never (score of 0)" to "Always (score of 4)
FreBAQ score in a subgroup of 50 subjects (35 patients and 15 controls) | Day 7
  a 9-item self-administered questionnaire, each item measured on a 5-point Likert scale ranging from "Never (score of 0)" to "Always (score of 4)
Evaluation of the internal consistency of the French version of the FreBAQ | Day 0
  Analyzed by calculating Cronbach's alpha.
Evaluation of the unidimensionality of the French version of the FreBAQ | Day 0
  Analyzed using principal component analysis methods
Assessment of the reliability (test-retest) of the questionnaire in French | Day 7
  Measurement of the reliability of the questionnaire in French between the initial test and a test at Day 7: calculation of Bland & Altman's limits of agreement,
Assessment of the reproducibility (test-retest) of the questionnaire in French | Day 7
  Measurement of the reproducibility of the questionnaire in French between the initial test and a test at Day 7: calculation of the intra-class correlation coefficient
Assessment of the discriminant validity of the questionnaire in French | Day 0
  Comparison of scores between control subjects and chronic low back pain patients by calculating the area under the ROC curve
Assessment of the concurrent validity | Day 0
  Correlation of the French questionnaire score with the duration of low back pain
Correlation of the French questionnaire score with lumbar visual analog scale (VAS) at rest | Day 0
  FreBAQ score compared with VAS result
Correlation of the French questionnaire score with lumbar VAS in movement | Day 0
  FreBAQ score compared with VAS result
Correlation of the French questionnaire score with disability | Day 0
  FreBAQ score compared with Oswestry Disability Index - a 10-section questionnaire with a results calculated as a percentage
Correlation of the French questionnaire score with false beliefs | Day 0
  FreBAQ score compared with back beliefs questionnaire - a 14-tem questionnaire on a 0-5 scale
Correlation of the French questionnaire score with fear avoidance beliefs | Day 0
  FreBAQ score compared with Fear Avoidance Belief Questionnaire - 16-item questionnaire scored between 0-6. Scale 1 = beliefs about work with a score ranging from 0 -42; Scale 2 = beliefs about physical activity with a score ranging from 0-24
Correlation of the French questionnaire score with kinesiophobia | Day 0
  FreBAQ score compared with Tampa scale of Kinesiophobia - total score 68, with a cut-off of 40 for significant kinesiophobia
Correlation of the French questionnaire score with catastrophism | Day 0
  FreBAQ score compared with Pain Catastrophizing Scale - a 13-item questionnaire on a 0-4 Likert scale
Correlation of the French questionnaire score with anxiety and depression | Day 0
  FreBAQ score compared with Hospital Anxiety and Depression Scale - a 14-item questionnaire on a 0-9 Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Homs, Principal Investigator — CHU Nîmes
Locations (1):
- CHU de Nîmes, Nîmes, France

REFERENCES:
- [Result] Homs AF, Ragon A, Mura T, Terribile G, Alonso S, Dupeyron AF. Validation of the French version of the Fremantle Back Awareness Questionnaire in patients with chronic low back pain. Eur J Phys Rehabil Med. 2025 Apr;61(2):295-304. doi: 10.23736/S1973-9087.24.08412-0. Epub 2025 Mar 10. PMID 40066561